CLINICAL TRIAL: NCT01245491
Title: The Effects of Vibration on Hypoxia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institute of Aviation Medicine, Oslo, Norway (Other Government)
Responsible Party: Anthony S. Wagstaff, Institute of Aviation Medicine
Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: REK-2010/2021b
Record Dates: First submitted 2010-11-19; First posted 2010-11-22 (Estimated); Last update posted 2011-01-14 (Estimated); Status verified 2011-01

CONDITIONS: Hypoxia
MeSH Terms: conditions — Hypoxia | interventions — Vibration

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: Vibration — Whole-body vibration, 17 Hz, 1.1ms-2

SUMMARY:
The purpose of this study is:

1. To study the effect of whole-body vibration on partial pressure of oxygen in arterial blood (PaO2), under hypobaric hypoxic conditions.
2. To study the effects of whole-body vibration and hypobaric hypoxia on visual contrast sensitivity.
3. To se if there is an increase in cytokines and other biomarkers under different hypobaric hypoxic conditions Our main hypothesis is that whole-body vibration may cause PaO2 to drop to a lower level, at a given altitude; than would be the case if there were no vibration present.

ELIGIBILITY:
Inclusion Criteria:

Exclusion Criteria:

* Stay at altitude over 2000 m last two weeks prior to study-start.
* Severe head injury
* Cardiovascular disease
* lung disease
* Decompression sickness

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2010-10; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
PaO2 | 14 minutes
  Assessed at six different altitudes
PaO2 | 35 minutes
  Assessed at six dfferent altitudes

SECONDARY OUTCOMES:
Ventilation | 14 minutes
  Assessed at six different altitudes, over a period of three minutes.
Ventilation | 35 minutes
  Assessed over a periode of three minutes, at six different altitudes.

CONTACTS AND LOCATIONS:
Overall Officials: Tor A Hansen, Msc., Principal Investigator — Institute of Aviation Medicine